CLINICAL TRIAL: NCT02867215
Title: Whole Barley Bread: Effect on the Risk of Metabolic Disease and Other Health Effects
Brief Title: Barley Bread and Metabolic Disease
Acronym: Barleybread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-15010303
Record Dates: First submitted 2016-07-19; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Barley bread (Active Comparator): Two loaves, 2 x 120 g loaf/day for 3 weeks.
  Interventions: Other: Barley bread
- Wheat bread (Active Comparator): Two loaves, 2 x 120 g loaf/day for 3 weeks.
  Interventions: Other: Wheat bread

INTERVENTIONS:
Other: Barley bread — 120g barley bread per day for 3 weeks.
  Arms: Barley bread
Other: Wheat bread — 120g wheat bread per day for 3 weeks.
  Arms: Wheat bread

SUMMARY:
The aim of this study was to compare the metabolic effects of consuming whole barley bread and whole wheat bread, in healthy subjects. Also, to investigate the effect of whole grain flour on mineral status.

DETAILED DESCRIPTION:
Generally, diet can be improved in order to lower diet-related diseases risk. However, the increasing prevalence rates of diet-related diseases indicate that, in practice, people's diet does not follow the recommendations. The intake of whole flour foods is consistently associated with reduced risk of type 2 diabetes and cardiovascular diseases in epidemiological studies, although the mechanisms of this association are unclear. Here the aim is to compare the metabolic effects and mineral status of consumption of diet containing wholemeal barley bread versus whole meal wheat bread in healthy subjects.

The intervention was designed as a randomized, cross over trial of 3-weeks duration. A total of 14 participants was included in the study. In one period subjects received WBB bread; in the second period, subjects received WWB bread. This bread is based on the recipe of Egyptian Baladi bread but formed in Danish buns form. Participants incorporated this bread into their normal habitual diet with regard to the study restrictions about other cereal food products. At the beginning and end of each intervention period blood was drawn and urine collected and stored for later analysis.

The primary outcomes of this study are evaluation of LDL-c, insulin and glucose levels evaluated by analysis of fasting blood samples. Furthermore, selected measures to evaluate SCFA level in blood is to be evaluated. Secondary outcomes include mineral status.

ELIGIBILITY:
Inclusion Criteria:

* Like and tolerate wheat/ barley bread products.
* Age: 20 - 53 years
* Body mass index (BMI): 23 - 30 kg/m2
* Weight stable (<3 kg weight change during the last 6 months)
* Apparently healthy
* Informed consent signed
* Freezer capacity for 1 week bread provision
* Can attend all visits required for the study

Exclusion Criteria:

* Wheat/gluten or barley intolerance
* Smoking on a daily basis
* Lactating (or lactating within 6 weeks prior to study start), pregnant (or pregnant within 3 months prior to study start) or wish to become pregnant during the study
* Diagnosed with any form of diabetes or cardiovascular disease
* Reported chronic gastrointestinal disorders
* Taking dietary supplements during or one month prior to the study
* Lack of cooperation and adherence to the protocol
* Use of prescription medication will be evaluated on an individual basis
* Blood donation within 3 months prior to study start or during the study
* Participation in other clinical trials

Ages: 20 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
LDL-c levels evaluated by analysis of fasting blood samples | 8-9 weeks
  Evaluated by analysis of fasting blood samples
Glucose levels evaluated by analysis of fasting blood samples | 8-9 weeks
  Evaluated by analysis of fasting blood samples
Insulin levels evaluated by analysis of fasting blood samples | 8-9 weeks
  Evaluated by analysis of fasting blood samples

SECONDARY OUTCOMES:
Mineral status | 8-9 weeks
  Evaluation depends on the mineral. Either by Atom absorption, ICP-MS or spectrometry

IPD SHARING:
Plan to Share IPD: Yes